CLINICAL TRIAL: NCT04048629
Title: Impact of Point-of-Care (POC) Viral Load (VL) Testing on Ensuring Appropriate Management of Viremia During Pregnancy to Prevent Vertical Transmission: an Observational Difference-in-difference Cohort Study
Brief Title: Impact of Point-of-care (POC) Viral Load (VL) Testing During Pregnancy in Zimbabwe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinton Health Access Initiative Inc. (Other)
Collaborators: Ministry of Health and Child Welfare, Zimbabwe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: POC VL during pregnancy
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: HIV Infections
Keywords: Zimbabwe; HIV; Viral load; Point-of-care; GeneXpert
MeSH Terms: conditions — HIV Infections | interventions — Surgical Instruments; Viral Load

STUDY DESIGN:
Intervention Model Description: This study is an observational cohort study with a baseline assessment, which will be used to conduct a difference in difference (DiD) analysis. The study design allows for assessment in more than one cross-section: 1) intervention clusters will be compared with control and 2) post-intervention clusters will be compared with an earlier baseline condition in control and intervention arms. The intervention (POC compared to centralized VL) is being offered at the facility level, as viral load testing is an intervention that is carried out on a clinic level, rather than at an individual patient level. The study is intended to investigate the effect of offering on-site POC VL testing on the proportion of enrolled PWLHIV who are virally suppressed at the time of delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point-of-care (POC) (Experimental): All facilities will receive a refresher training on Zimbabwe's 2018 Guidelines. At POC facilities, at the first antenatal visit (ANC1), all women enrolled in the intervention cohort will have a blood sample collected for VL which will be tested onsite using an existing POC device. If a woman is virally unsuppressed (VL ≥1000 cpm), she will be given adherence counseling and, if necessary, a treatment regimen switch/infant prophylaxis per national guidelines.
  Interventions: Device: Point-of-care (POC) viral load (VL) testing plus refresher training
- Standard of care (SOC) (Active Comparator): All facilities will receive a refresher training on Zimbabwe's 2018 Guidelines. At SOC facilities, at ANC1, all women enrolled in the intervention cohort will have a blood sample collected for VL which will be sent to centralized labs for testing. If a woman is virally unsuppressed (VL ≥1000 cpm), she will be given adherence counseling and, if necessary, a treatment regimen switch/infant prophylaxis per national guidelines.
  Interventions: Other: Standard of care central laboratory VL testing plus refresher training

INTERVENTIONS:
Device: Point-of-care (POC) viral load (VL) testing plus refresher training — VL testing at the first antenatal care visit will occur using POC VL testing in pregnant women, and a refresher training on Zimbabwe's guidelines will be provided at all facilities
  Other Names: GeneXpert
  Arms: Point-of-care (POC)
Other: Standard of care central laboratory VL testing plus refresher training — VL testing at the first antenatal care visit will occur using central laboratory VL testing in pregnant women, and a refresher training on Zimbabwe's guidelines will be provided at all facilities
  Arms: Standard of care (SOC)

SUMMARY:
The Ministry of Health and Child Care (MOHCC) in collaboration with Clinton Health Access Initiative (CHAI) will conduct an observational cohort study to determine the impact and cost-effectiveness of POC VL testing for pregnant women. It is hypothesized that POC VL testing will enable an increased proportion of pregnant women to be virally suppressed at delivery, which will avert vertical transmission.

DETAILED DESCRIPTION:
Twenty public health facilities that offer HIV care to pregnant women and maternity services will be included in the study with half offering VL testing at the first antenatal care visit using the centralized VL system (standard of care cluster) and the other half offering onsite POC VL (POC cluster). The primary end-point will be the proportion of enrolled pregnant women who are virally suppressed at the time of delivery. Positivity rate will be measured as a secondary outcome. Primary and secondary outcomes will be compared between study arms. As well, a baseline assessment in each facility will be included to enable a difference in difference analysis within clusters, in which viral suppression rates at delivery and other outcomes are compared before and after the intervention.

The primary research question to be addressed by this study is: Does the availability of POC VL testing during ANC increase the proportion of women who are virally suppressed at the time of delivery?

The primary objective is to demonstrate the impact of POC VL on ensuring viral suppression at the time of delivery (defined as a viral load < 1,000 cpm within 2 weeks of delivery) for pregnant women living with HIV (PWLHIV) who are on ART in order to avert vertical transmission.

In addition, this study will:

* document the at-birth and 4-6 week EID positivity rate
* document proportion of women who have undetectable VL at the time of delivery (defined as below the limit of detection (LOD) of the VL test)
* document the baseline coverage of VL monitoring during the first ANC visit for WLHIV on ART ≥ 6 months
* compare the timeliness of VL result receipt by clinics (HCW) and clients between facilities with POC VL and those using centralized testing
* calculate the cost-effectiveness of POC VL for increasing the proportion of women who are virally suppressed at delivery

ELIGIBILITY:
Sites will be selected for inclusion in the study based on following criteria:

* Offer HIV testing and antiretroviral therapy (ART) services
* Offer prevention of mother-to-child transmission (PMTCT) and maternity services
* Offer Viral load monitoring either using POC or through referral
* Availability of Second line ART
* Located in 2 provinces in which VL testing labs are located
* Have historic monthly ANC cohorts of ≥ 6 pregnant women living with HIV (PWLHIV) already on ART

Patient Inclusion Criteria:

Baseline Cohort:

All women living with HIV on ART ≥7 months who deliver at the study facilities during the enrollment period, who do not meet the study criteria for the intervention cohort, were on ART at ANC1 and are of the age of consent (≥ 18 years old) will be offered participation. Informed consent will be obtained to collect a study-specific blood sample to perform a VL test in the central lab at the time of delivery. 7 months has been selected to be comparable to women in the intervention cohort who may present for ANC1 at 4 weeks prior to delivery who are on ART ≥ 6 months.

Intervention Cohort:

Pregnant women who are known to be living with HIV and on ART for ≥ 6 months and attend the study facilities for ANC services and have an anticipated due date ≥ 4 weeks, will be offered participation in the study. It is expected that a woman who is on ART < 6 months may not yet have achieved viral suppression (using current NNRTI-containing regimens) and therefore conducting a VL at this time is not currently standard. According to Zimbabwe guidelines and consistent with normative guidance from the World Health Organization (WHO), any infant born to a woman living with HIV who is on ART for less than 4 weeks is considered at high risk of HIV transmission. Therefore, for this study the first ANC visit must be ≥ 4 weeks prior to delivery. Women must be at least the age of adult consent (≥ 18 years old) in Zimbabwe. If consent is obtained, a sample will be collected at ANC1 for VL testing.

Patient Exclusion Criteria:

Baseline Cohort

* PWLHIV not on ART at ANC1 or on ART < 7 months at time of delivery
* Women who have enrolled in or are eligible for the intervention cohort
* Women who are not HIV positive
* Pregnant women who are newly diagnosed as HIV positive during pregnancy
* Women who cannot or do not provide informed consent

Intervention Cohort

* Pregnant women who are newly diagnosed as HIV positive during pregnancy
* PWLHIV not on ART or on ART < 6 months at their first ANC visit
* Women who are not HIV positive
* Women who cannot or do not provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1715 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Viral suppression at delivery | Within 2 weeks after delivery
  The proportion of enrolled PWLHIV on ART ≥ 6 months at their first ANC visit who are virally suppressed at delivery

SECONDARY OUTCOMES:
Viral suppression at delivery among those with an unsuppressed viral load at first antenatal care visit | Within 2 weeks after delivery
  The proportion of enrolled PWLHIV identified as having unsuppressed VL at first ANC who suppress at delivery
Infant HIV infection | Within 6 weeks of birth
  The proportion of infants who test HIV positive at birth and/or 4-6 weeks using an early infant diagnosis (EID) test
Turnaround time to VL results available at facility | Through end of the study, approximately 1 year
  The time between VL sample collection and result receipt by health care provider
Turnaround time to VL results available to patient | Through end of the study, approximately 1 year
  The time between VL sample collection and result receipt by pregnant woman living with HIV

OTHER OUTCOMES:
Costing of POC VL | Through end of the study, approximately 1 year
  The commodity costs of VL testing at ANC1 on the POC platform will be calculated ($USD per patient) and compared to the commodity costs of VL testing using the central laboratory given any differences in the primary and secondary endpoints by group
Acceptability of POC VL | End of the study, approximately 1 year after study start
  The acceptability to healthcare workers of offering POC VL testing at the first ANC visit, based on a survey

CONTACTS AND LOCATIONS:
Locations (20):
- Zimbabwe (20):
  - Luveve Clinic, Bulawayo
  - Mpilo Central Hospital, Bulawayo
  - Nkulumane Clinic, Bulawayo
  - Pelandaba Clinic, Bulawayo
  - United Bulawayo Hospital, Bulawayo
  - Budiriro PolyClinic, Harare
  - Chitungwiza Central Hospital, Harare
  - Gleview, Harare
  - Hatcliffe PolyClinic, Harare
  - Highfield PolyClinic, Harare
  - Kambuzuma, Harare
  - Kuwadzana PolyClinic, Harare
  - Mabvuku PolyClinic, Harare
  - Mbare PolyClinic, Harare
  - Rujeko, Harare
  - Rutsanana PolyClinic, Harare
  - Seke South Clinic, Harare
  - St. Mary's Clinic, Harare
  - Warren Park PolyClinic, Harare
  - Zengeza Clinic, Harare

IPD SHARING:
Plan to Share IPD: No